CLINICAL TRIAL: NCT07080970
Title: Observational Study on APL-like Subset Within NPM1-mutated Acute Myeloid Leukemia: a Distinct Phenotypic Signature Correlating With Early-onset Vascular Complications. ACTIVATE (APL-like aCute Myeloid Leukemia: disTInct Phenotype and Early VAscular complicaTions)
Brief Title: Observational Study on APL-like aCute Myeloid Leukemia: disTInct Phenotype and Early VAscular complicaTions
Acronym: ACTIVATE
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: AML3025
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; NPM1 Mutation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APL-like: NPM1 AML patients identified as APL-like cohort
  Interventions: Other: observation of incidence of early vascular events
- Non APL-like: NPM1 AML patients identified as no APL-like cohort
  Interventions: Other: observation of incidence of early vascular events

INTERVENTIONS:
Other: observation of incidence of early vascular events — observation of difference incidence of early vascular events in the two cohorts

SUMMARY:
This is a multicenter observational study with a retrospective and a prospective cohort investigating clinically and biologically the APL-like subset as a potential predictor of coagulopathy and susceptibility to early vascular events.

DETAILED DESCRIPTION:
This is a multicenter observational study with a retrospective and a prospective cohort investigating clinically and biologically the APL-like subset as a potential predictor of coagulopathy and susceptibility to early vascular events.

Participating Centers will identify NPM1-mutated patients eligible for enrollment. The immune-phenotypic data will be evaluated to define a specific signature to be applied for the identification of APL-like AML.

All patients will be followed for a minimum of 12 months until the study closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with de novo AML, untreated, newly diagnosed, according to WHO/ICC 2022 criteria from January 2015 onwards.
* Presence of NPM1 mutation.
* Availability of immunophenotypic characterization at diagnosis
* Age >= 18 years
* Signed written informed consent according to ICH/EU/GCP and national local laws (if applicable)

Exclusion Criteria:

* No specific exclusion criteria are provided once eligibility criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will include NPM1mut AML patients with an immunophenotypic characterization at diagnosis that allows the classification into APL-like and non-APL-like AML.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of early vascular events | 30 days from diagnosis
  Evaluation of the incidence of early vascular events (haemorrhagic and/or thrombotic) in the APL-like and non-APL-like subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Mannelli, Principal Investigator — SOD Ematologia, Università di Firenze, AOU Careggi